CLINICAL TRIAL: NCT01602666
Title: Phase 2 Trial of Response-Based Radiation Therapy for Patients With Localized Central Nervous System Germ Cell Tumors (CNS GCT)
Brief Title: Chemotherapy Followed by Radiation Therapy in Treating Younger Patients With Newly Diagnosed Localized Central Nervous System Germ Cell Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACNS1123; NCI-2012-01967 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000734032; S12-02807; ACNS1123 (Other: Children's Oncology Group); ACNS1123 (Other: CTEP); K12CA086913 (NIH); U10CA098543 (NIH); U10CA180886 (NIH)
Record Dates: First submitted 2012-05-18; First posted 2012-05-21 (Estimated); Results first posted 2020-12-16 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Central Nervous System Nongerminomatous Germ Cell Tumor; Childhood Germinoma
MeSH Terms: interventions — Radiotherapy, Conformal; Carboplatin; Etoposide; Ifosfamide; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (combination chemotherapy, radiation therapy) (Experimental): See Detailed Description
  Interventions: Radiation: 3-Dimensional Conformal Radiation Therapy; Drug: Carboplatin; Drug: Etoposide; Drug: Ifosfamide; Radiation: Intensity-Modulated Radiation Therapy

INTERVENTIONS:
Radiation: 3-Dimensional Conformal Radiation Therapy — Undergo 3D-CRT
  Other Names: 3-dimensional radiation therapy; 3D Conformal; 3D CONFORMAL RADIATION THERAPY; 3D CRT; 3D radiotherapy; 3D-CRT; Conformal Therapy; Radiation Conformal Therapy; Radiation, 3D Conformal; Three dimensional external beam radiation therapy (procedure)
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; JM8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16; VP 16-213; VP 16213; VP-16; VP-16-213; VP-16213; VP16; VP16213
Drug: Ifosfamide — Given IV
  Other Names: Asta Z 4942; Asta Z-4942; Cyfos; Holoxan; Holoxane; Ifex; IFO; IFO-Cell; Ifolem; Ifomida; Ifomide; Ifosfamidum; Ifoxan; IFX; Iphosphamid; Iphosphamide; Iso-Endoxan; Isoendoxan; Isophosphamide; Mitoxana; MJF 9325; MJF-9325; Naxamide; Seromida; Tronoxal; Z 4942; Z-4942
Radiation: Intensity-Modulated Radiation Therapy — Undergo IMRT
  Other Names: IMRT; Intensity modulated radiation therapy (procedure); Intensity Modulated RT; Intensity-Modulated Radiotherapy; Radiation, Intensity-Modulated Radiotherapy

SUMMARY:
This phase II trial studies how well chemotherapy followed by radiation therapy work in treating younger patients with newly diagnosed central nervous system germ cell tumors that have not spread to other parts of the brain, spinal canal, or body (localized). Drugs used as chemotherapy, such as carboplatin, etoposide, and ifosfamide, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Radiation therapy uses high-energy x rays to kill tumor cells. Giving chemotherapy followed by radiation therapy may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine, as measured by the 3-year progression-free survival (PFS) rate and patterns of failure, whether dose and volume of irradiation can be safely reduced to 30.6 Gy whole ventricular-field irradiation (WVI) plus 23.4 Gy primary site boost instead of 36 Gy craniospinal irradiation (CSI) plus primary site boost in the subgroup of children and young adults (ages 3 to =< 21 years) with localized nongerminomatous germ cell tumor (NGGCT) who have a magnetic resonance imaging (MRI) and tumor marker criteria (cerebrospinal fluid [CSF] and serum) for confirmed complete response (CR) or partial response (PR) to induction chemotherapy and negative serum and cerebrospinal fluid (CSF) tumor markers OR in patients who have less than a PR after induction chemotherapy with negative tumor markers who undergo a second-look surgery and are found to have only mature teratoma, residual scar or fibrosis and fit the definition of CR/PR after second-look surgery.

II. To determine, as measured by the 3-year PFS rate and patterns of failure, whether simplified chemotherapy followed by dose-reduced radiation therapy is effective for treating children and young adults (ages 3 to =< 21 years) with localized primary central nervous system (CNS) germinoma who present with serum and/or CSF human chorionic gonadotropin-beta (hCGbeta) =< 50 mIU/mL.

III. To prospectively evaluate and longitudinally model the cognitive, social, and behavioral functioning of children and young adults who are treated with reduced radiation dose and volume of irradiation in Stratum 1 (NGGCT) and with dose-reduced radiation therapy in Stratum 2 (germinoma) using the ALTE07C1 protocol.

SECONDARY OBJECTIVES:

I. To estimate the PFS and overall survival (OS) distributions of patients with NGGCT treated with 30.6 Gy WVI and involved-field radiation therapy (IFR) focal boost to 54 Gy.

II. To estimate the PFS and OS distributions of localized germinoma patients who present with a) serum and/or CSF hCGbeta =< 50 mIU/mL and b) serum and/or CSF hCGbeta > 50 mIU/mL and =< 100 mIU/mL.

OUTLINE:

STRATUM I (NGGCT): Patients receive induction therapy comprising carboplatin intravenously (IV) over 15-60 minutes on day 1 and etoposide IV over 60-120 minutes on days 1-3 of courses 1, 3, and 5. Patients also receive ifosfamide IV over 60 minutes and etoposide over 60-120 minutes on days 1-5 of courses 2, 4, and 6. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity. Patients achieving CR or PR undergo 3-dimensional conformal radiation therapy (3DRT) or intensity modulated radiation therapy (IMRT) once daily (QD) 5 days a week for 6 weeks. Patients with normalization of markers who fail to achieve CR or PR are strongly recommended to undergo second-look surgery. Patients who achieve CR or PR after second-look surgery undergo 3DRT or IMRT QD 5 days a week for 6 weeks.

STRATUM II (GERMINOMA): Patients receive induction therapy comprising carboplatin IV over 15-60 minutes on day 1 and etoposide IV over 60-120 minutes on days 1-3. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity. Patients with CR or continued CR (CCR) undergo 3DRT or IMRT QD 5 days a week for 4 weeks. Patients with normalization of markers who fail to achieve CR or PR are strongly recommended to undergo second-look surgery. Patients found to have fibrosis, scar, mature teratoma, or non-viable tumor undergo 3DRT or IMRT QD 5 days a week for 4 weeks. Patients with stable disease (SD) or PR with > 0.5 cm (suprasellar) or > 1 cm (pineal) but =< 1.5 cm residual disease do not undergo second-look surgery and undergo 3DRT or IMRT QD 5 days a week for 4 weeks.

After completion of study treatment, patients are followed up at 3, 6, and 9 months, every 4 months for 24 months, 30 months, 36 months, and then annually for up to 60 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be newly diagnosed with localized primary CNS NGGCT (Stratum 1) or localized primary CNS germinoma (Stratum 2); germ cell tumors located in the suprasellar, pineal, bifocal (pineal + suprasellar) and ventricles are eligible; tumors present in the above mentioned locations and with unifocal parenchymal extension are eligible

  * Stratum 1(NGGCT): Patients must have one of the following criteria:

    * Patients with serum and/or CSF hCGbeta > 100 mIU/mL or any elevation of serum and/or CSF alpha-fetoprotein (AFP) > 10 ng/mL or greater than the institutional normal are eligible, irrespective of biopsy results
    * Patients with any of the following elements on biopsy/resection are eligible, irrespective of serum and/or CSF hCGbeta and AFP levels: endodermal sinus tumor (yolk sac), embryonal carcinoma, choriocarcinoma, malignant/immature teratoma, and mixed GCT with malignant GCT elements
  * Stratum 2 (Germinoma): Patients must have both serum and CSF markers obtained (unless obtaining CSF is medically contraindicated) and must have one of the following criteria to be eligible:

    * Patients with institutional normal AFP (or =< 10 ng/mL if no institutional normal exists) in both serum and CSF (unless medically contraindicated) AND hCGbeta 5 to =< 50 mIU/mL in serum and/or CSF (unless medically contraindicated) (only 1 is required to be elevated) are eligible; no histologic confirmation required
    * Patients with bifocal (pineal + suprasellar) involvement or pineal lesion with diabetes insipidus (D1) AND hCGbeta =< 100 mIU/mL in serum and/or CSF AND institutional normal AFP (or =< 10 ng/mL if no institutional normal exists) in both serum and CSF (unless medically contraindicated) are eligible; no histologic confirmation required
    * Patients with histologically confirmed germinoma or germinoma mixed with mature teratoma and hCGbeta =< 100 mIU/mL in serum and/or CSF and institutional normal AFP (or =< 10 ng/mL if no institutional normal exists) in both serum and CSF (unless medically contraindicated) are eligible
* All patients must have a cranial MRI with and without gadolinium at diagnosis/prior to enrollment; if surgical resection is performed, patients must have pre-operative and post-operative cranial MRI with and without gadolinium; the post-operative brain MRI should be obtained within 72 hours of surgery; if patient has a biopsy only, post-operative cranial MRI is recommended but not required; all patients must have a spine MRI with gadolinium obtained at diagnosis/prior to enrollment; Note: if the spine study is performed for the first time after surgical resection or biopsy, it is recommended to be obtained with and without gadolinium
* Lumbar CSF must be obtained prior to study enrollment unless medically contraindicated; if a patient undergoes surgery and lumbar CSF cannot be obtained at this time, then it should be performed at least 10 days following surgery before study enrollment; false positive cytology can occur within 10 days of surgery; Note: patients with positive CSF cytology obtained prior to 10 days after surgery may have cytology repeated to determine eligibility
* Patients must have CSF tumor markers obtained prior to enrollment unless medically contraindicated; ventricular CSF obtained at the time of CSF diversion procedure (if performed) is acceptable for tumor markers but lumbar CSF is preferred; in case CSF diversion and biopsy/surgery are combined, CSF tumor markers should be collected first
* Patients must be enrolled on ALTE07C1 prior to enrollment on ACNS1123; patients must be enrolled within 31 days of definitive diagnostic surgery (day 0) or clinical diagnosis
* Peripheral absolute neutrophil count (ANC) >= 1,000/uL
* Platelet count >= 100,000/uL (transfusion independent)
* Hemoglobin >= 8.0 g/dL (may receive red blood cell [RBC] transfusions)
* Creatinine clearance or radioisotope glomular filtration rate (GFR) >= 70 mL/min/1.73 m^2 OR serum creatinine based on age/gender as follows:

  * 0.8 mg/dL (2 to < 6 years of age)
  * 1.0 mg/dL (6 to < 10 years of age)
  * 1.2 mg/dL (10 to < 13 years of age)
  * 1.5 mg/dL (male) and 1.4 mg/dL (female) (13 to < 16 years of age)
  * 1.7 mg/dL (male) and 1.4 mg/dL (female) (>= 16 years of age)
* Total bilirubin =< 1.5 times upper limit of normal (ULN) for age
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) and serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) < 2.5 times ULN
* Patients with seizure disorder may be enrolled if well controlled
* Patients must not be in status, coma, or assisted ventilation prior to study enrollment

Exclusion Criteria:

* Patients with mature teratoma or completely resected immature teratoma with normal tumor markers are not eligible
* Patients with tumors located outside the ventricles (basal ganglia, thalamus) are not eligible
* Patients with metastatic disease by cranial or spinal MRI evaluation or CSF cytology (unless medically contraindicated) are not eligible
* Patients must not have received any prior tumor-directed therapy other than surgical intervention and corticosteroids
* Female patients who are pregnant are ineligible
* Lactating females are not eligible unless they have agreed not to breastfeed their infants
* Female patients of childbearing potential are not eligible unless a negative pregnancy test result has been obtained
* Sexually active patients of reproductive potential are not eligible unless they have agreed to use an effective contraceptive method for the duration of their study participation
* All patients and/or their parents or legal guardians must sign a written informed consent
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 262 (Actual)
Dates: Start 2012-06-27 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ute K Bartels, Principal Investigator — Children's Oncology Group
Locations (167):
- United States (149):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Kaiser Permanente Downey Medical Center, Downey, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Mattel Children's Hospital UCLA, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center, Torrance, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Lee Memorial Health System, Fort Myers, Florida
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Clinic - Orlando, Orlando, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Tampa General Hospital, Tampa, Florida
  - Saint Mary's Medical Center, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Advocate Children's Hospital-Oak Lawn, Oak Lawn, Illinois
  - Advocate Children's Hospital-Park Ridge, Park Ridge, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Michigan State University, East Lansing, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Albany Medical Center, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Mission Hospital, Asheville, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Greenville Cancer Treatment Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - T C Thompson Children's Hospital, Chattanooga, Tennessee
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - UMC Cancer Center / UMC Health System, Lubbock, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Carilion Children's, Roanoke, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Australia (9):
  - John Hunter Children's Hospital, Hunter Regional Mail Centre, New South Wales
  - Sydney Children's Hospital, Randwick, New South Wales
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Royal Children's Hospital-Brisbane, Herston, Queensland
  - Queensland Children's Hospital, South Brisbane, Queensland
  - Women's and Children's Hospital-Adelaide, North Adelaide, South Australia
  - Royal Children's Hospital, Parkville, Victoria
  - Princess Margaret Hospital for Children, Perth, Western Australia
  - Perth Children's Hospital, Perth, Western Australia
- Canada (6):
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
- New Zealand (2):
  - Starship Children's Hospital, Grafton, Auckland
  - Christchurch Hospital, Christchurch
- University Pediatric Hospital, San Juan, Puerto Rico

REFERENCES:
- [Derived] Fangusaro J, Wu S, MacDonald S, Murphy E, Shaw D, Bartels U, Khatua S, Souweidane M, Lu HM, Morris D, Panigrahy A, Onar-Thomas A, Fouladi M, Gajjar A, Dhall G. Phase II Trial of Response-Based Radiation Therapy for Patients With Localized CNS Nongerminomatous Germ Cell Tumors: A Children's Oncology Group Study. J Clin Oncol. 2019 Dec 1;37(34):3283-3290. doi: 10.1200/JCO.19.00701. Epub 2019 Sep 23. PMID 31545689

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients enrolled on the study from 6/27/2012 to 11/1/2016 on Stratum 1 and from 6/27/2012 to 10/26/2018 on Stratum 2
Pre-assignment Details: There were 111 patients enrolled in Stratum 1 with localized nongerminomatous germ cell tumors (NGGCT) and 151 patients enrolled in Stratum 2 with localized CNS Germinoma (Germinoma). Of these 107 in Stratum 1 and 137 in Stratum 2 were deemed eligible for the study. This report is limited to eligible subjects.
Groups:
- Stratum 1 Localized Non-Germinomatous Germ Cell Tumors (NGGCT): Patients receive induction therapy comprising carboplatin intravenously (IV) over 15-60 minutes on day 1 and etoposide IV over 60-120 minutes on days 1-3 of courses 1, 3, and 5. Patients also receive ifosfamide IV over 60 minutes and etoposide over 60-120 minutes on days 1-5 of courses 2, 4, and 6. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity. Patients achieving CR or PR undergo 3-dimensional conformal radiation therapy (3DRT) or intensity modulated radiation therapy (IMRT) once daily (QD) 5 days a week for 6 weeks. Patients with normalization of markers who fail to achieve CR or PR are strongly recommended to undergo second-look surgery. Patients who achieve CR or PR after second-look surgery undergo 3DRT or IMRT QD 5 days a week for 6 weeks.
- Stratum 2 Localized Germinoma: Patients receive induction therapy comprising carboplatin IV over 15-60 minutes on day 1 and etoposide IV over 60-120 minutes on days 1-3. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity. Patients with CR or continued CR (CCR) undergo 3DRT or IMRT QD 5 days a week for 4 weeks. Patients with normalization of markers who fail to achieve CR or PR are strongly recommended to undergo second-look surgery. Patients found to have fibrosis, scar, mature teratoma, or non-viable tumor undergo 3DRT or IMRT QD 5 days a week for 4 weeks. Patients with stable disease (SD) or PR with > 0.5 cm (suprasellar) or > 1 cm (pineal) but =< 1.5 cm residual disease do not undergo second-look surgery and undergo 3DRT or IMRT QD 5 days a week for 4 weeks.
Period: Induction Chemotherapy
Arm/Group | Stratum 1 Localized Non-Germinomatous Germ Cell Tumors (NGGCT) | Stratum 2 Localized Germinoma
Started | 107 | 137
Completed | 70 | 113
Not Completed | 37 | 24
Not completed — Death | 2 | 1
Not completed — Lack of Efficacy | 16 | 7
Not completed — Physician Decision | 12 | 5
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Refusal of further protocol therapy | 5 | 6
Not completed — Radiotherapy can't be initiated in 6 wks | 2 | 3
Period: Radiation Therapy on Protocol
Arm/Group | Stratum 1 Localized Non-Germinomatous Germ Cell Tumors (NGGCT) | Stratum 2 Localized Germinoma
Started | 70 | 113
Evaluable for Reduced Dose (30Gy) | 66 | 0
Evaluable for Reduced Dose (18 Gy) | 0 | 74
Evaluable for RT Dose (24Gy) | 0 | 16
Completed | 60 | 82
Not Completed | 10 | 31
Not completed — Lost to Follow-up | 4 | 5
Not completed — Withdrawal by Subject | 2 | 3
Not completed — In-evaluable for reduced dose(30.6 Gy) | 4 | 0
Not completed — In-evaluable for reduced dose(18 Gy) | 0 | 14
Not completed — In-evaluable for RT dose (24Gy) | 0 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stratum 1 Localized Non-Germinomatous Germ Cell Tumors (NGGCT) | Stratum 2 Localized Germinoma | Total
Number analyzed (Participants) | 107 | 137 | 244
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 100 | 124 | 224
  Between 18 and 65 years | 7 | 13 | 20
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 11.0 [3.7 to 21.6] | 14.1 [5.0 to 21.5] | 13.0 [3.7 to 21.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 37 | 64
  Male | 80 | 100 | 180
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 16 | 36
  Not Hispanic or Latino | 83 | 113 | 196
  Unknown or Not Reported | 4 | 8 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 8 | 14 | 22
  Native Hawaiian or Other Pacific Islander | 1 | 8 | 9
  Black or African American | 6 | 9 | 15
  White | 78 | 86 | 164
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 14 | 19 | 33
Region of Enrollment [Number; unit: participants]
  United States | 93 | 117 | 210
  Australia | 7 | 10 | 17
  Canada | 7 | 6 | 13
  New Zealand | 0 | 4 | 4

OUTCOME MEASURES:

1. Primary Outcome: 3-year Progression-free Survival (PFS) Rate of Patients With Nongerminomatous Germ Cell Tumor (NGGCT) Who Were Treated With Reduced Dose Whole Ventricular-field Irradiation
Description: Binomial estimate of the 3-year PFS rate defined as "Yes" for patients who were followed up per protocol and were progression free at 3-years, and "No" for those who either experienced a progression or were lost to follow-up/withdrew from the trial within 3 years from enrollment. Progression was determined by MRI using the COG Guidelines for Measurement of Tumor Size (>25% increase in 2D or >40% in 3D of the product of perpendicular diameters of the target lesion) as well as by tumor marker assessments which were mandatory for this study.
Time Frame: 3 years
Population: Localized NGGCT treated with 30.6 Gy WVF RT + 23.4 Gy primary site boost. Patients must have had complete response (CR) or partial response (PR) to induction chemotherapy by MRI and markers; or underwent second-look surgery and were found to have mature teratoma, residual scar or fibrosis and fit the definition of CR/PR after second-look surgery.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Stratum 1 Localized Non-Germinomatous Germ Cell Tumors (NGGCT)
Number analyzed (Participants) | 66
percentage of patients | 83.33 [72.13 to 91.38]

2. Primary Outcome: 3-year PFS Rate of Patients With Localized CNS Germinoma Who Were Treated With Reduced Dose Radiation Therapy
Description: Binomial estimate of the 3-year PFS rate defined as "Yes" for patients who were followed up per protocol and were progression free at 3-years, and "No" for those who either experienced a progression or were lost to follow-up/withdrew from the trial within 3 years from initiation of treatment. Progression was determined by MRI using the COG Guidelines for Measurement of Tumor Size (>25% increase in 2D or >40% in 3D of the product of perpendicular diameters of the target lesion) as well as by tumor marker assessments which were mandatory for this study.
Time Frame: 3 years
Population: Localized CNS Germinoma treated with dose-reduced RT (18 Gy WVI + 12 Gy primary site boost) and had complete response (CR) after induction chemotherapy by MRI and tumor marker criteria; or underwent second-look surgery and were found to have mature teratoma, residual scar or fibrosis and fit the definition of CR after second-look surgery.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Stratum 2 Localized Germinoma
Number analyzed (Participants) | 74
percentage of patients | 86.49 [76.55 to 93.32]

3. Primary Outcome: Neurocognitive Function Using the ALTE07C1 Protocol
Description: Estimated scores for the cognitive functions of processing speed, attention/concentration, and estimated IQ were assessed using the age-appropriate version of the Wechsler Scales of Intelligence. The range for the Processing Speed Index (PSI) is 45 to 155, with a mean of 100 and a standard deviation of 15. Estimated IQ was estimated using 2 subtests from the Wechsler Scales of Intelligence to derive a standard score with a mean of 100 and standard deviation of 15 with a range of 45 to 158. Scores from the 2 subtests were summed and translated to a standard score using published procedures. Attention/concentration was measured by the Digit Span subtest score from the Wechsler Scales of Intelligence. Subset scores have a range of 1-19, with a mean of 10 and standard deviation of 3. Higher scores on all these measures indicate higher or better cognitive performance, lower scores indicate lower or worse cognitive functioning.
Time Frame: Up to 5 years
Population: All eligible patients who received the radiation therapy were included as evaluable patients for analysis.
Measure: Mean (95% Confidence Interval); unit: Standardized Scores
Arm/Group | Stratum 1 Localized Non-Germinomatous Germ Cell Tumors (NGGCT) | Stratum 2 Localized Germinoma
Number analyzed (Participants) | 70 | 113
Standardized Scores
  Attention/Concentration at 9 months: number analyzed (Participants) | 50 | 85
  Attention/Concentration at 9 months | 9.4 [8.6 to 10.3] | 10.0 [9.3 to 10.7]
  Attention/Concentration at 30 months: number analyzed (Participants) | 40 | 69
  Attention/Concentration at 30 months | 10.1 [9.1 to 11.1] | 9.8 [9.0 to 10.6]
  Attention/Concentration at 60 months: number analyzed (Participants) | 28 | 44
  Attention/Concentration at 60 months | 9.3 [8.3 to 10.4] | 10.2 [9.1 to 11.3]
  Estimated IQ at 9 months: number analyzed (Participants) | 48 | 94
  Estimated IQ at 9 months | 94.3 [90.0 to 98.7] | 99.0 [95.9 to 102.1]
  Estimated IQ at 30 months: number analyzed (Participants) | 44 | 72
  Estimated IQ at 30 months | 101.3 [96.2 to 106.4] | 102.9 [99.1 to 106.7]
  Estimated IQ at 60 months: number analyzed (Participants) | 29 | 45
  Estimated IQ at 60 months | 97.3 [91.2 to 103.5] | 104.5 [100.0 to 108.9]
  Processing Speed at 9 months: number analyzed (Participants) | 48 | 94
  Processing Speed at 9 months | 90.1 [85.2 to 94.9] | 91.8 [88.3 to 95.3]
  Processing Speed at 30 months: number analyzed (Participants) | 44 | 70
  Processing Speed at 30 months | 93.4 [87.7 to 99.0] | 95.6 [92.3 to 98.9]
  Processing Speed at 60 months: number analyzed (Participants) | 29 | 45
  Processing Speed at 60 months | 90.1 [82.2 to 98.0] | 97.5 [93.1 to 101.9]

4. Secondary Outcome: Estimation of the PFS Distribution of Patients With NGGCT Treated With Involved-field Radiation Therapy (IFR)
Description: Kaplan Meier estimate of the 3-year PFS is provided. PFS is the time interval measured from enrollment until progression or death from any cause or until last follow-up for those who were event free at the time of analysis. Patients who were lost to follow-up or withdrew consent were censored in this analysis. Progression was determined by MRI using the COG Guidelines for Measurement of Tumor Size (>25% increase in 2D or >40% in 3D of the product of perpendicular diameters of the target lesion) as well as by tumor marker assessments which were mandatory for this study.
Time Frame: Up to 3 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Stratum 1 Localized Non-Germinomatous Germ Cell Tumors (NGGCT)
Number analyzed (Participants) | 66
percentage of patients | 87.88 [77.22 to 93.75]

5. Secondary Outcome: Estimation of the Overall Survival (OS) Distribution of Patients With NGGCT Treated With IFR Assessed
Description: Kaplan Meier estimate of the 3-year overall survival (OS) is provided. OS is the time interval measured from enrollment until death from any cause or until last follow-up for those who were alive at the time of analysis. Patients who were lost to follow-up or withdrew consent were censored in this analysis.
Time Frame: Up to 3 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Stratum 1 Localized Non-Germinomatous Germ Cell Tumors (NGGCT)
Number analyzed (Participants) | 66
percentage of patients | 92.42 [82.75 to 96.78]

6. Secondary Outcome: Estimation of the PFS Distribution of Patients With Localized Germinoma Patients and Cerebrospinal Fluid (CSF) Serum hCGbeta of 50 mIU/mL or Less or CSF Serum hCGbeta Greater Than 50 mIU/mL and Less Than or Equal to 100 mIU/mL
Description: Kaplan Meier estimate of the 3-year PFS rate is provided. PFS is the time interval measured from initiation of treatment until progression or death from any cause or until last follow-up for those who were event free at the time of analysis. Patients who were lost to follow-up or withdrew consent were censored in this analysis. Progression was determined by MRI using the COG Guidelines for Measurement of Tumor Size (>25% increase in 2D or >40% in 3D of the product of perpendicular diameters of the target lesion) as well as by tumor marker assessments which were mandatory for this study.
Time Frame: Up to 3 years
Population: The eligible patients with localized germinoma and CSF serum hCGbeta of 50 mIU/mL or less or CSF serum hCGbeta greater than 50 mIU/mL and less than or equal to 100 mIU/mL.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Groups:
- hCGbeta <= 50 mIU/mL: CSF/serum hCGbeta <= 50 mIU/mL
- 50 mIU/mL < hCGbeta <= 100 mIU/mL: 50 mIU/mL < CSF /serum hCGbeta <= 100 mIU/mL
Arm/Group | hCGbeta <= 50 mIU/mL | 50 mIU/mL < hCGbeta <= 100 mIU/mL
Number analyzed (Participants) | 131 | 6
percentage of patients | 93.26 [86.95 to 96.58] | 80.00 [20.38 to 96.92]

7. Secondary Outcome: Estimation of the OS Distribution of Patients With Localized Germinoma Patients and CSF Serum hCGbeta of 50 mIU/mL or Less or CSF Serum hCGbeta Greater Than 50 mIU/mL and Less Than or Equal to 100 mIU/mL
Description: Kaplan Meier estimate of the 3-year overall survival (OS) is provided for each group. OS is the time interval measured from enrollment until death from any cause or until last follow-up for those who were alive at the time of analysis. Patients who were lost to follow-up or withdrew consent were censored in this analysis.
Time Frame: Up to 3 years
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | hCGbeta <= 50 mIU/mL | 50 mIU/mL < hCGbeta <= 100 mIU/mL
Number analyzed (Participants) | 131 | 6
percentage of patients | 98.38 [93.69 to 99.59] | 100 [100 to 100]

ADVERSE EVENTS:
Time Frame: From initiation of induction of therapy to the date of last follow-up, approximately 3 years. For most subjects the adverse events were observed while on active treatment or shortly thereafter.
Description: Adverse event reporting is collected routinely using case report forms. The SAE table reflects NCI Common Terminology Criteria for Adverse Events (CTCAEs) submitted by the institution via expedited reporting (NCI AdEERs / CAeRs). All remaining CTCAEs collected by means other than expedited reporting are non-serious and are reported in the "AE Other" table. Ineligible patients are excluded from reporting of adverse events. All-Cause Mortality includes all deaths collected on the study.
Arm/Group | Stratum 1 Localized Non-Germinomatous Germ Cell Tumors (NGGCT) | Stratum 2 Localized Germinoma
All-Cause Mortality (participants affected / at risk) | 13/107 | 2/137
Serious Adverse Events (participants affected / at risk) | 5/107 | 1/137
Other Adverse Events (participants affected / at risk) | 84/107 | 107/137
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stratum 1 Localized Non-Germinomatous Germ Cell Tumors (NGGCT) (N=107) | Stratum 2 Localized Germinoma (N=137)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stratum 1 Localized Non-Germinomatous Germ Cell Tumors (NGGCT) (N=107) | Stratum 2 Localized Germinoma (N=137)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 2 (2)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 10 (13) | 15 (23)
Allergic reaction (Immune system disorders) | 0 (0) | 3 (3)
Anal mucositis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anaphylaxis (Immune system disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 45 (99) | 48 (101)
Anorexia (Metabolism and nutrition disorders) | 6 (7) | 2 (2)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0)
Avascular necrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Blood and lymphatic system disorders - Other- Specify (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 2 (2) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
CPK increased (Investigations) | 1 (1) | 0 (0)
Catheter related infection (Infections and infestations) | 3 (4) | 0 (0)
Cerebrospinal fluid leakage (Nervous system disorders) | 1 (1) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 3 (3) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 6 (7) | 8 (10)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 4 (4) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dysphasia (Nervous system disorders) | 1 (1) | 0 (0)
Edema cerebral (Nervous system disorders) | 0 (0) | 1 (1)
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 5 (5) | 0 (0)
Endocrine disorders - Other- Specify (Endocrine disorders) | 0 (0) | 2 (2)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Eye pain (Eye disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 19 (28) | 22 (31)
GGT increased (Investigations) | 1 (3) | 1 (1)
Growth suppression (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 7 (8) | 2 (2)
Hearing impaired (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hydrocephalus (Nervous system disorders) | 5 (6) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (4) | 4 (5)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypernatremia (Metabolism and nutrition disorders) | 18 (33) | 14 (15)
Hypersomnia (Nervous system disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 11 (17) | 15 (19)
Hyponatremia (Metabolism and nutrition disorders) | 23 (32) | 14 (21)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2) | 5 (7)
Hypotension (Vascular disorders) | 3 (3) | 1 (1)
Hypothermia (General disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
INR increased (Investigations) | 1 (1) | 0 (0)
Infections and infestations - Other- Specify (Infections and infestations) | 3 (7) | 1 (1)
Infusion related reaction (General disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Intracranial hemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Irritability (General disorders) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 2 (2) | 1 (1)
Lymph gland infection (Infections and infestations) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 31 (85) | 11 (12)
Lymphocyte count increased (Investigations) | 0 (0) | 1 (1)
Mania (Psychiatric disorders) | 1 (1) | 0 (0)
Meningismus (Nervous system disorders) | 1 (1) | 0 (0)
Mucosal infection (Infections and infestations) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Multi-organ failure (General disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 4 (5)
Neoplasms benign- malignant and unspecified (incl cysts and polyps) - Other- Specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 0 (0)
Nervous system disorders - Other- Specify (Nervous system disorders) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 66 (210) | 92 (266)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0)
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 54 (126) | 83 (213)
Renal and urinary disorders - Other- Specify (Renal and urinary disorders) | 1 (1) | 1 (1)
Seizure (Nervous system disorders) | 2 (2) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 2 (2)
Somnolence (Nervous system disorders) | 3 (4) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 3 (4)
Thromboembolic event (Vascular disorders) | 3 (3) | 0 (0)
Upper respiratory infection (Infections and infestations) | 3 (3) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 7 (8) | 6 (9)
Weight gain (Investigations) | 1 (1) | 1 (1)
White blood cell decreased (Investigations) | 52 (150) | 50 (88)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior approval

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-06-01): https://cdn.clinicaltrials.gov/large-docs/66/NCT01602666/Prot_SAP_000.pdf